CLINICAL TRIAL: NCT01496469
Title: A Phase 2, Double-Blind, Placebo-Controlled Study to Assess the Effect of Febuxostat 80 mg Once Daily Compared to Placebo on Ambulatory Blood Pressure in Subjects With Hyperuricemia and Hypertension
Brief Title: Effect of Febuxostat on Blood Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMX-67_206; U1111-1124-4638 (Registry Identifier: WHO)
Record Dates: First submitted 2011-12-18; First posted 2011-12-21 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-07

CONDITIONS: Hypertension
Keywords: Drug Therapy
MeSH Terms: conditions — Hypertension | interventions — Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Febuxostat 80 mg QD (Experimental): Febuxostat 80 mg, tablets, orally, once daily for up to 6 weeks.
  Interventions: Drug: Febuxostat
- Placebo QD (Placebo Comparator): Febuxostat placebo-matching tablets, orally, once daily for up to 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Febuxostat — Febuxostat 80 mg, tablets, orally, once daily for up to 6 weeks
  Other Names: TMX-67; Uloric
  Arms: Febuxostat 80 mg QD
Drug: Placebo — Febuxostat placebo-matching tablets, orally, once daily for up to 6 weeks.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to evaluate the effect of febuxostat, once daily (QD), compared to placebo on lowering ambulatory 24-hour mean blood pressure of participants with hypertension and hyperuricemia (not associated with gout).

DETAILED DESCRIPTION:
This study is designed to evaluate the effect of febuxostat during 6 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The participant has documented hypertension, defined as average clinic systolic blood pressure (SBP) of ≥145 mm Hg and ≤165 mm Hg or average clinic diastolic blood pressure (DBP) of ≥90 mm Hg and ≤105 mm Hg at the Day -21 Screening Visit; the average BP measurement at two of the three Placebo Run-in Visits (Day -14, Day -7 and Day -1) must also meet the above criteria for hypertension.
2. The participant has a serum uric acid (sUA) level ≥7.0 mg/dL not associated with gout, at the Day -21 Screening Visit.
3. The participant has a 24-hour mean ambulatory SBP of ≥130 mm Hg and < 165 mm Hg at the Baseline (Day 1) Visit.
4. At the initial Screening Visit (Day -21), the maximum number of antihypertensive medications the participant is taking is ≤ 2 (fixed-dose combination medications are considered 2 medications, including diuretics), and the participant has been on a stable dose of this medication for at least1 month prior to start of the initial Screening Visit (Day -21).
5. The participant is male and at least 18 years of age, or a female who is:

   * Surgically sterilized (hysterectomy, bilateral oophorectomy or tubal ligation), OR
   * Postmenopausal (defined as at least 1 year since last regular menses with an follicle-stimulating hormone (FSH) >40 IU/L, or at least 5 years since last regular menses), OR
   * On hormone replacement therapy and ≥ 55 years of age.
6. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
7. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.

Exclusion Criteria:

1. The participant has received any investigational compound within 30 days, or within 5 half-lives of the compound (whichever is longer) prior to the Screening Visit.
2. The participant has received febuxostat or any urate-lowering therapy (ULT) in a previous clinical study or as a therapeutic agent.
3. The participant has gout, history of gout, or gout flares.
4. The participant has secondary hyperuricemia (HPU) (e.g., due to myeloproliferative disorder, or organ transplant).
5. The participant has known secondary hypertension of any etiology (e.g., renovascular disease, primary hyperaldosteronism, Cushing syndrome).
6. The participant has a history, within the 6 months prior to screening, of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, or percutaneous coronary intervention.
7. The participant has an irregular cardiac rhythm (e.g., atrial fibrillation, multifocal premature atrial contractions) which leads to difficulty with interpretation of ambulatory blood pressure monitoring (ABPM).
8. The participant has a history of congestive heart failure, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack.
9. The participant has type 1 or poorly controlled type 2 diabetes mellitus (glycosylated hemoglobin [HbA1c] >8.0%) at Screening.
10. The participant has a history of infection with hepatitis B, hepatitis C, or human immunodeficiency virus.
11. The participant has an average clinic SBP >165 mm Hg or DBP >105 mm Hg at 1 or more visits during the Placebo Run-in Period.
12. The participant's average clinic SBP or DBP measurement that increases or decreases by >10 mm Hg between Placebo Run-in visits (Day -14 to Day -7, or Day -7 to Day -1, or Day -14 to Day -1).
13. The participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.
14. The participant has an alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) values greater than 2.0 times the upper limit of normal (ULN).
15. The participant has a significant medical condition and/or conditions that would interfere with the treatment, safety or compliance with the protocol.
16. The participant has a history of alcoholism or illicit drug abuse within 5 years prior to the Screening Visit or is currently consuming >14 alcoholic drinks per week.
17. The participant has a known hypersensitivity or allergies to febuxostat or any components of the formulations of this compound.
18. The participant is taking or expected to take a medication as described in the excluded medication section.
19. The participant has a history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug. This criterion does not apply to those participants with successfully resected basal cell or stage I squamous cell carcinoma of the skin.
20. The participant's estimated glomerular filtration rate (eGFR) is <30 mL/min/1.73m3, where eGFR is calculated by the Central Laboratory using the Modification of Diet in Renal Disease (MDRD) formula at the Day -21 Screening Visit.
21. The participant is noncompliant (<80% or >120%) with study medication during Placebo Run-In Period.
22. The participant has an upper arm circumference less than 24 cm or greater than 42 cm.
23. The participant's work shift includes any hour between 11 PM (2300) to 7 AM (0700).
24. The participant has a baseline 24-hour ABPM reading of insufficient quality (as described in Appendix F of the protocol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (45):
- United States (45):
  - Foley, Alabama
  - Buena Park, California
  - Carmichael, California
  - Fresno, California
  - Irvine, California
  - Lomita, California
  - Paramount, California
  - Sacramento, California
  - San Diego, California
  - Wildomar, California
  - Milford, Connecticut
  - Fort Lauderdale, Florida
  - Miami, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Dunwoody, Georgia
  - Roswell, Georgia
  - Suwanee, Georgia
  - Avon, Indiana
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Biddeford, Maine
  - City of Saint Peters, Missouri
  - St Louis, Missouri
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Glens Falls, New York
  - Greensboro, North Carolina
  - Salisbury, North Carolina
  - Shelby, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Lyndhurst, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Tipton, Pennsylvania
  - Carrollton, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Burke, Virginia
  - Manassas, Virginia
  - Port Orchard, Washington
  - Madison, Wisconsin

REFERENCES:
- [Derived] Gunawardhana L, McLean L, Punzi HA, Hunt B, Palmer RN, Whelton A, Feig DI. Effect of Febuxostat on Ambulatory Blood Pressure in Subjects With Hyperuricemia and Hypertension: A Phase 2 Randomized Placebo-Controlled Study. J Am Heart Assoc. 2017 Nov 4;6(11):e006683. doi: 10.1161/JAHA.117.006683. PMID 29102979
- See also: Uloric Package Insert — http://general.takedapharm.com/content/file.aspx?applicationcode=6C7C39D8-5D09-453B-BF30-696A4AB88E62&fileTypeCode=ULORICPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 29 sites in the United States from 10 January 2012 to 04 August 2014.
Pre-assignment Details: Participants with a historical diagnosis of hypertension along with hyperuricemia were enrolled in 1 of 2 treatment groups as follows: Placebo; Febuxostat 80 milligram (mg).
Groups:
- Placebo: Febuxostat placebo-matching over-encapsulated tablet, orally, once daily for up to 6 weeks.
- Febuxostat 80 mg: Febuxostat 80 mg, over-encapsulated tablet, orally, once daily for up to 6 week.
Period: Overall Study
Arm/Group | Placebo | Febuxostat 80 mg
Started | 60 | 61
Completed | 50 | 53
Not Completed | 10 | 8
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 4 | 4
Not completed — BP exceeds protocol limits | 1 | 2
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants who were randomized and received at least 1 dose of double-blind study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Febuxostat 80 mg | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.08 (10.607) | 52.15 (10.469) | 53.60 (10.597)
Age, Customized [Number; unit: participants]
  Less than (<) 45 years | 8 | 14 | 22
  45 - <65 years | 44 | 43 | 87
  Greater than or equal to (>=) 65 years | 8 | 4 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 48 | 50 | 98
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 7 | 8 | 15
  Black or African American | 11 | 10 | 21
  White | 42 | 41 | 83
  More than one race | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 9 | 14 | 23
  Not Hispanic or Latino | 51 | 47 | 98
Region of Enrollment [Number; unit: participants]
  United States | 60 | 61 | 121
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 172.10 (8.564) | 173.33 (9.206) | 172.72 (8.878)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 95.35 (21.199) | 100.88 (19.490) | 98.14 (20.460)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 31.99 (5.133) | 33.55 (5.913) | 32.78 (5.572)
BMI Category [Number; unit: participants]
  18.5 - <25 | 3 | 3 | 6
  25 - <30 | 18 | 17 | 35
  >=30 | 39 | 41 | 80
Smoking History [Number; unit: participants]
  Never smoked | 32 | 30 | 62
  Current smoker | 8 | 10 | 18
  Ex-smoker | 20 | 21 | 41
Alcohol History [Number; unit: participants]
  Never Drunk | 26 | 20 | 46
  Current Drinker | 32 | 37 | 69
  Ex-Drinker | 2 | 4 | 6
Renal Function [Number; unit: participants] — Renal function categories were defined by estimated glomerular filtration rate (eGFR) calculated based on modification of diet in renal disease (MDRD) formula. Moderately impaired = eGFR 30 to 59 milliliter per minute (mL/min); mildly impaired = eGFR 60 to 89 mL/min; normal renal function=eGFR >=90 mL/min.
  participants
    Moderately Impaired | 8 | 5 | 13
    Mildly Impaired | 33 | 30 | 63
    Normal | 19 | 26 | 45
Baseline serum uric acid (sUA) [Number; unit: participants]
  < 8.0 milligram per deciliter (mg/dL) | 40 | 47 | 87
  >=8.0 mg/dL | 20 | 14 | 34
Baseline Medication [Number; unit: participants] — Baseline medication included angiotensin receptor blocker (ARB) and angiotensin-converting enzyme inhibitors (ACEi).
  participants
    ARB or ACEi | 26 | 28 | 54
    None | 34 | 33 | 67

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-hour Mean Systolic Blood Pressure (SBP) Measured by Ambulatory Blood Pressure Monitoring at Week 6
Description: The change in 24-hour mean SBP measured at final visit or Week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 6
Population: FAS included all participants who were randomized and received at least 1 dose of double-blind study medication and had a baseline value and at least 1 post-baseline value available, with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | Febuxostat 80 mg
Number analyzed (Participants) | 53 | 56
millimeters of mercury (mmHg)
  Baseline | 142.3 (1.21) | 139.5 (1.18)
  Change at Week 6 | -3.4 (1.31) | -3.7 (1.27)
Statistical Analysis 1: Comparison: Placebo vs Febuxostat 80 mg; A total of 120 enrolled participants (60 participants per treatment group) was sufficient to achieve 80 percent (%) power to detect a difference of 6.0 mmHg between the placebo and febuxostat 80 mg treatment groups by a 2 sample t-test of the mean change from Baseline at Week 6 in 24-hour mean ambulatory SBP with a 2-sided significance level of 5%; Test type: Superiority or Other; p = 0.882, ANCOVA — Analysis of covariance (ANCOVA) model with treatment as a factor, and the baseline value and prior use of an ARB or an ACEi as covariates; Least Squares Mean Difference = -0.3, 95% CI 2-sided [-3.9 to 3.4]

2. Secondary Outcome: Change From Baseline in 24-hour Mean Diastolic Blood Pressure (DBP) Measured by Ambulatory Blood Pressure Monitoring at Week 6
Description: The change in 24-hour mean DBP measured at final visit or Week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Febuxostat 80 mg
Number analyzed (Participants) | 53 | 56
mmHg
  Baseline | 85.9 (1.14) | 83.0 (1.11)
  Change at Week 6 | -2.7 (0.91) | -2.0 (0.88)
Statistical Analysis 1: Comparison: Placebo vs Febuxostat 80 mg; ANCOVA model with treatment as a factor, and the baseline value and prior use of an ARB or an ACEi as covariates; Test type: Superiority or Other; p = 0.613, ANCOVA — Tested at 5% significance level; Least Squares Mean Difference = 0.6, 95% CI 2-sided [-1.9 to 3.2]

3. Secondary Outcome: Change From Baseline in Serum Urate Levels at Week 6
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Febuxostat 80 mg
Number analyzed (Participants) | 52 | 51
mg/dL
  Baseline | 7.7 (0.14) | 7.6 (0.14)
  Change at Week 6 | 0.1 (0.17) | -3.3 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Febuxostat 80 mg; ANCOVA model with treatment as a factor, and the baseline value and prior use of an ARB or an ACEi as covariates; Test type: Superiority or Other; p < 0.001, ANCOVA — Tested at 5% significance level; Least Squares Mean Difference = -3.4, 95% CI 2-sided [-3.9 to -2.9]

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs are defined as any AEs, regardless of relationship to study drug, which occurs on or after the first double-blind dose date and up to 30 days after the last dose date of the double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Febuxostat 80 mg
Serious Adverse Events (participants affected / at risk) | 1/60 | 1/61
Other Adverse Events (participants affected / at risk) | 1/60 | 3/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=60) | Febuxostat 80 mg (N=61)
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=60) | Febuxostat 80 mg (N=61)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.